CLINICAL TRIAL: NCT03480815
Title: Nocturnal Temperature Controlled Laminar Airflow Device, Airsonett, for Treating Severe Allergic Asthma After Withdrawal of Omalizumab therapyT
Brief Title: Nocturnal TLA for Severe Allergic Asthma After Withdrawal of Omalizumab Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Principal Investigator, Chun-Hua Wang, MD, Professor, MD, Chang Gung Memorial Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 201600573A3
Record Dates: First submitted 2018-03-05; First posted 2018-03-29 (Actual); Last update posted 2021-06-09 (Actual); Status verified 2018-03

CONDITIONS: Severe Allergic Asthma
Keywords: Asthma; Controlled Laminar Airflow Device; Omalizumab
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Intervention Model Description: a randomized, controlled study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TLA device (Active Comparator): These patients will be withdrawal of omalizumab treatment and receive nocturnal temperature controlled laminar flow device at nighttime for 12 months.
  Interventions: Device: Nocturnal Temperature Controlled Laminar Flow Device
- None device (Placebo Comparator): These patients will be withdrawal of omalizumab treatment and do not receive TLA device for 12 months.
  Interventions: Other: None Device

INTERVENTIONS:
Device: Nocturnal Temperature Controlled Laminar Flow Device — Record of the time to first asthma exacerbation, lung function and exhaled NO level
  Arms: TLA device
Other: None Device — Record of the time to first asthma exacerbation, lung function and exhaled NO level
  Arms: None device

SUMMARY:
This is a randomized, controlled study with a 48-week treatment phase to determine the clinical efficacy of temperature controlled laminar flow device (TLA, Airsonett™) in the patients with severe allergic asthma who are withdrawal of omalizumab therapy

DETAILED DESCRIPTION:
This is a randomized, controlled study with a 48-week treatment phase to determine the clinical efficacy of temperature controlled laminar flow device (TLA, Airsonett™) in the patients with severe allergic asthma who are withdrawal of omalizumab therapy. All patients will be recruited from outpatient clinics of Thoracic Department of Chang Gung Memorial Hospital and meet the inclusion criteria. After entry the study, these patients will continuous their concomitant asthma medicines, except the treatment of omalizumab. These patients will be randomized (1:1) to receive TLA device or matching Control group. The participants will be recorded by randomized number to protect their private information. To minimize a potential treatment group imbalance of clinical asthma management practice and concomitant asthma medication use, randomization will be stratified by concomitant asthma medication [in addition to inhaled corticosteroid (ICS) and long-acting β2-agonist (LABA)] use at baseline: (1) patients not receiving theophylline, oral β2-agonists, antileukotrienes or maintenance oral steroids; (2) patients receiving one or more from theophylline, oral β2-agonists and anti-leukotrienes, but not receiving maintenance oral steroids; (3) patients receiving maintenance oral steroids. The doses of ICS and LABA (taken separately or as a fixed combination) and other concomitant asthma medications will be kept constant through the treatment period. If they have asthma exacerbation of emergency visit or/and hospitalization, or > or =2 episodes of asthma exacerbation (defined as a worsening of asthma symptoms requiring treatment with systemic corticosteroids), the patients either with TLA or Control group will return to start the omalizumab therapy till the end of 48-week follow-up. Omalizumab dose is based on the patient's body weight and total serum immunoglobulin E (IgE) level at screening and is administered every 2 or 4 weeks to provide a dose of at least 0.016 mg/kg per IU/ml of IgE. Patients are permitted short-acting β2-agonist rescue medication as required.

Patients make study visits at weeks 0, 2, 4, 12, 24, 36 and 48 of the treatment phase. The primary efficacy variable is the first time to asthma exacerbations during the 48-week TLA treatment phase. Rate of hospitalization, and emergency visit per year will be also recorded. Diary cards are used to record the clinical symptom score, asthma control test (ACT) and use of rescue medication in the internet of Asthma Help.

Quality of life will be assessed using the Sino-Nasal Outcome Test (SNOT-22) score at weeks 0, 12, 24, 36 and 48 of the treatment phase. Spirometry and exhaled NO will be performed at each visit. All visits include assessment of vital signs and physical examination.

ELIGIBILITY:
Inclusion Criteria:

1. Willing to sign a written consent form
2. Male and female subjects were diagnosed severe allergic asthma and received omalizumab as add-on therapy for more 4 than months and had stable asthma control.
3. Men and women over the age of 20 and less than 80 year-old
4. Accept application of TLA or not after withdrawal of omalizumab therapy
5. Positive reaction of specific IgE (Phadiatop) for one or more than on indoor allergens.

Exclusion Criteria:

1. Having an exacerbation within 4 weeks before entry the study
2. Using immunosuppressants within 3 months of the first visit
3. Having recent upper airway infection or systemic corticosteroid usage within 4 weeks
4. Bronchiectasis
5. Active pulmonary tuberculsis
6. COPD
7. Cystic fibrosis

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2017-01-20 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
The first time of asthma exacerbation | Through study completion of 48 weeks
  Time to the first significant asthma exacerbation or ER visit or hospitalization will be also recorded.

SECONDARY OUTCOMES:
Spirometry | at 0, 4, 12, 24, 36, and 48 weeks after enrollment
  Pulmonary function testing, including FVC and FEV1
Exhaled nitric oxide | at 0, 4, 12, 24, 36, and 48 weeks after enrollment
  measured level is ppb.

CONTACTS AND LOCATIONS:
Overall Officials: Chun-Hua Wang, MD, Principal Investigator — Department of Thoracic Medicine, Chang Gung Memorial Hospital
Locations (1):
- Chang Gung Memorial Hospital, Taoyuan District, Taiwan

IPD SHARING:
Plan to Share IPD: No
N/D